CLINICAL TRIAL: NCT01882673
Title: Brief Computer Intervention to Motivate Quitline Use for Smokers in SUD Treatment
Brief Title: Motivating Quitline Use Among Smokers in Treatment for Substance Use Disorders
Acronym: MI-SUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA034312
Record Dates: First submitted 2013-06-10; First posted 2013-06-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Smoking Cessation
Keywords: Tobacco; nicotine; dependence; quitline
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Computer Motivational Interviewing for Smoking Cessation (Experimental): Brief computer motivational interviewing intervention to motivate tobacco quitline use
  Interventions: Behavioral: Brief Computer Motivational Interviewing for Smoking Cessation
- Nutrition Control (Active Comparator): Computer delivered nutrition education
  Interventions: Behavioral: Nutrition Control

INTERVENTIONS:
Behavioral: Brief Computer Motivational Interviewing for Smoking Cessation — Brief computer motivational interviewing intervention to motivated tobacco quitline use
  Arms: Brief Computer Motivational Interviewing for Smoking Cessation
Behavioral: Nutrition Control — Computer delivered nutrition education control condition
  Arms: Nutrition Control

SUMMARY:
The long-term goal of this program of research is to disseminate an effective, brief computer-based intervention that can be readily integrated into Substance Use Disorders (SUD) treatment programs to motivate tobacco quitline use in patients who smoke. The overall objective of this application, which is the first step in the attainment of this long-term goal, is to fully develop this computer-based intervention, modify it based on initial piloting and feedback to insure its feasibility and acceptability, and obtain preliminary data supporting the efficacy of the intervention. This will be accomplished by pursuing three specific aims: 1) to develop and conduct preliminary pilot testing (n=20) of a brief, computer-based intervention intended to motivate tobacco quitline use among cigarette smokers in SUD treatment (TIME-TQ; Tablet computer Intervention to Motivate Engagement in Tobacco Quitline use) and to develop and pilot test a computer-based, time matched control intervention (CON), 2) to conduct a preliminary randomized controlled trial (RCT) with 60 smokers in SUD treatment, comparing TIME-TQ vs. CON, with predictions that TIME-TQ relative to CON will result in increased readiness, higher rates of tobacco treatment engagement, more quit smoking attempts and higher rates of 7-day point prevalence abstinence rates at 1- and 3-month follow-ups. Substance use outcomes over the course of the 3-month follow-up period will also be examined, and 3) to examine TIME-TQ's effects on key mechanisms during the computer session and their associations with tobacco treatment engagement and smoking outcomes at 1- and 3-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 70 years of age
* current smoker (i.e., at least 10 cigarettes per day)
* current DSM-IV alcohol or drug abuse or dependence per SCID-P.

Exclusion Criteria:

* history of psychotic disorder or current psychotic symptoms per the Structured Clinical Interview for DSM 4R - Patient version
* cognitive impair-ment sufficient to impair provision of informed consent or study participation
* current suicidality or homicidality
* use of NRT or other pharmacotherapy for smoking cessation
* use of other tobacco products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Engaged in tobacco cessation treatment since end of treatment intervention | 3-months

SECONDARY OUTCOMES:
Number of quit smoking attempts since last assessment | 3-months

OTHER OUTCOMES:
Point prevalence smoking abstinence - last 7 days from time of assessment | 3-months

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Brown, Ph.D., Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States